CLINICAL TRIAL: NCT00431028
Title: Phase I/II Comparative Study of a Single Intraoperative Sub-Tenon's Capsule Injection of Triamcinolone and Ciprofloxacin in a Controlled-Release System Versus 1% Prednisolone and 0.3% Ciprofloxacin Eyedrops for Cataract Surgery
Brief Title: Sub-Tenon's Injection of Triamcinolone and Ciprofloxacin in a Controlled-Release System for Cataract Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated
Sponsor: Federal University of São Paulo (Other)
Responsible Party: fernando paganelli, federal university of sao paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Duocat 001
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Inflammation; Bacterial Infections
Keywords: Cataract; Endophthalmitis; Antibiotics; Anti-Inflammatory Agents; Drug Delivery Systems
MeSH Terms: conditions — Inflammation; Bacterial Infections; Cataract; Endophthalmitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- colirio (No Intervention): prednisolone 1% eye drops + ciprofloxacin 0,3% eye drops
  Interventions: Device: slow delivery ciprofloxacin + triamcinolone

INTERVENTIONS:
Device: slow delivery ciprofloxacin + triamcinolone — 2 mg ciprofloxacin + 25mg triamcinolone
  Other Names: ciprofloxacin; triamcinolona

SUMMARY:
The purpose of this study is to compare one intraoperative sub-Tenon's capsule injection of triamcinolone and ciprofloxacin in a biodegradable controlled-release system with conventional prednisolone and ciprofloxacin eye drops to treat ocular inflammation and for infection prophylaxis after cataract surgery.

DETAILED DESCRIPTION:
Topical steroids effectively control ocular inflammation, but are associated with the well-recognized problems of patient compliance. Injection of depot corticosteroids into sub-Tenon's capsule is an established method of treating various ocular inflammatory diseases. Its prolonged therapeutic effect has provided the ophthalmologist with an alternative tool for the treatment of different diseases that may be extended to the surgical arena to modulate postoperative inflammation.

The use of topical antibiotic agents poses unique and challenging hurdles for drug delivery, especially because recent reports have suggested that the incidence of endophthalmitis may be increasing. Exploiting the permeability of the sclera, subconjunctival routes may offer a more promising alternative for enhanced drug delivery and tissue targeting compared with topical routes. In theory, the combination of an antibiotic with a steroid in a controlled-release system delivered transscleral could be feasible after cataract surgery to achieve several clinical objectives, i.e., eliminate topical medications, enhance patient compliance, improve drug bioavailability, and protect the patient from infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncomplicated, senile cataract
* Best-corrected visual acuity (VA) of 20/100 or better in the fellow eye

Exclusion Criteria:

* Patients in use of oral or topical anti-inflammatory agents
* History of steroid-induced ocular hypertension
* Hypermature cataracts
* Previous ocular surgery
* Preexisting uveitis
* Diabetic retinopathy
* Glaucoma
* Corneal disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Anterior chamber cell | Days 1, 3, 7, 14, and 28 after surgery
Anterior chamber flare | Days 1, 3, 7, 14, and 28 after surgery
Intraocular pressure | Days 1, 3, 7, 14, and 28 after surgery
Lack of anti-inflammatory response | Days 1, 3, 7, 14, and 28 after surgery
Presence of infection | Days 1, 3, 7, 14, and 28 after surgery

SECONDARY OUTCOMES:
Conjunctival hyperemia | Days 1, 3, 7, 14, and 28 after surgery
Spectacle corrected visual acuity | Day 28 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Paganelli, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Department of Ophthalmology, Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Paganelli F, Cardillo JA, Melo LA Jr, Lucena DR, Silva AA Jr, Oliveira AG, Hofling-Lima AL, Nguyen QD, Kuppermann BD, Belfort R Jr; Brazilian Ocular Pharmacology and Pharmaceutical Technology Research Group. A single intraoperative sub-tenon's capsule injection of triamcinolone and ciprofloxacin in a controlled-release system for cataract surgery. Invest Ophthalmol Vis Sci. 2009 Jul;50(7):3041-7. doi: 10.1167/iovs.08-2920. Epub 2009 Feb 21. PMID 19234342